CLINICAL TRIAL: NCT00263003
Title: A Randomized, Open Label Comparative Study of Irbesartan/Hydrochlorothiazide and Irbesartan in the Treatment of Mild to Moderate Hypertension
Brief Title: Irbesartan/Hydrochlorothiazide and Irbesartan in the Treatment of Mild to Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM_L_0094
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2007-12-07 (Estimated); Status verified 2007-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: Irbesartan/hydrochlorothiazide
Drug: Irbesartan

SUMMARY:
Study Objectives :

* To demonstrate the reduction in office Blood Pressure following a 8-week regimen of irbesartan / hydrochlorothiazide using irbesartan as a reference.
* To demonstrate the reduction in office Blood Pressure after 4-week regimen of irbesartan / hydrochlorothiazide using irbesartan as a reference.
* To compare the response rate (defined as office Systolic Blood Pressure/Diastolic Blood Pressure reduce more than 10mmHg from Week 0) of patients after 4-week and 8-week regimen of irbesartan / hydrochlorothiazide versus irbesartan.
* To compare the proportion of patients requiring titration after 4-week regimen of irbesartan/hydrochlorothiazide versus irbesartan
* To ascertain the safety and tolerability of irbesartan / hydrochlorothiazide versus irbesartan when administered once daily

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate hypertension with office Diastolic Blood Pressure (DBP) 90-109 mmHg and/or Systolic Blood Pressure (SBP) 140-179 mmHg
* All women of child-bearing potential must have negative urine pregnancy tests within a week prior to initiation of therapy

Exclusion Criteria:

* females who are pregnant or breast feeding
* office DBP ≥ 110 mmHg or office SBP ≥ 180 mmHg
* history of significant cardiovascular diseases which includes:

  * acute myocardial infarction within six months or any ischemic heart disease requiring medication.
  * cerebrovascular disease
* history of significant renal diseases including:

  * serum creatinine > 3.0 mg/dl.
  * creatinine clearance < 30 ml/min.
* severe biliary cirrhosis and cholestasis
* refractory hypokalemia, hypercalcemia
* history of autoimmune disease, collagen vascular disease, multiple drug allergies, bronchospastic disease or other malignancies requiring current medication
* hepatic disease as indicated by any of the following:

  * SGOT or SGPT >3 x upper limit of normal.
  * Serum bilirubin > 2 x upper limit of normal.
* any other condition or therapy that, in the investigator's opinion, or as indicated in the product(s) label may pose a risk to the patient or interfere with the study objectives.
* any other investigational drug given within 30 days of initiation of therapy, and participation in other clinical studies while enrolled in this protocol.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-06

PRIMARY OUTCOMES:
Compare the reduction in office BP following a 8-week regimen of irbesartan / hydrochlorothiazide versus irbesartan

SECONDARY OUTCOMES:
Compare the reduction in office BP following a 4-week regimen of irbesartan / hydrochlorothiazide versus irbesartan
Compare the response rate (defined as office SBP/DBP reduce more than 10mmHg from week 0) of patients after 4-week and 8-week regimen of irbesartan/hydrochlorothiazide versus irbesartan
Compare the proportion of patients requiring titration after 4-week regimen of irbesartan/hydrochlorothiazide versus irbesartan
Ascertain the safety and tolerability of irbesartan/hydrochlorothiazide versus irbesartan when administered once daily.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon CHANG, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Taipei, Taiwan